Page 1|2 Version: 2 | 12/23/2021

### TITLE OF RESEARCH: NEURAL CIRCUITRIES OF MOTOR LEARNING AS A TARGET TO MODULATE SENSORIMOTOR RECOVERY AFTER STROKE

### **Medical University of South Carolina**

## STANDARDIZED TEXT TO BE READ TO POTENTIAL PARTICIPANTS BEFORE THE TELEPHONE SCREENING

I am contacting you today to ask you to volunteer for a research study because you

# [a) is read to a potential volunteer for the stroke group, b) is read to a potential volunteer for the control group]

- a) have experienced a stroke at least six months ago and have been experiencing difficulties moving parts of your body or using your hand and arm in your daily activities since your stroke.
- **b)** have never experienced a stroke, and may be a participant in the control group.

Research studies are voluntary and include only people who choose to take part. The purpose of this study is to better understand how brain areas communicate with each other when a new movement skill is learned, and how this communication changes during the recovery of movement after stroke.

The investigator in charge of this study is Dr. Kirstin-Friederike Heise. This study is being performed at MUSC and will involve three visits over two weeks at the Stroke Recovery Research Center and the Center for Biomedical Imaging in Charleston.

If you decide to participate, we will ask you to complete an interview and computerized tests that assess your physical and mental health, medical, cognition, and mood history at your first visit. During the second and third visits, you will practice a task similar to playing a video game. During this task, you will learn how to adjust your grip force on a moving prompt that you can see on a computer screen. You will also receive MRI brain scans at both visits which will require you to lie on a long narrow bed while the machine gathers data.

There are risks, discomforts, and inconveniences associated with any research study. The possible risks associated with this study include possible emotional distress, pain or claustrophobia from the MRI machine and possible loss of confidentiality. There is no direct benefit for you from participating in this study. Participating in this study is completely voluntary and participation is not required.

If you have any more questions about participating in this study, you may contact Dr. Kirstin-Friederike Heise at (843) 792-3435.

To make sure that your participation in the study is safe for you and that you can take part in all parts of the study, I want to ask you some specific questions on the phone today. These questions involve a brief assessment of your cognitive function, for example your

IRB Number: «ID»

Date Approved «ApprovalDate»



Page 2|2 Version: 2 | 12/23/2021

ability to remember words or calculate.

[the following sentence is only read to a potential volunteer for the stroke group]

In addition, I will ask you about your ability to move your hand and arm that are most affected by the stroke.

#### [the following is read to all potential participants, stroke and controls]

This telephone interview will take 20-30 minutes to complete. If you agree to take part in this telephone interview, you will be given more detailed information about the study procedures afterwards and you will have time to decide if you want to participate in the study.

Only if you decide to participate in the study and sign the consent form, will we keep the information collected in this telephone interview. If you decide not to participate or if we find out that the participation would not be safe for you, we will destroy the information collected today.

Your participation in this study is entirely voluntary. The same is true for this telephone interview today. You may refuse to take part in or stop taking part in this interview at any time.

By participating in this telephone interview, you indicate that you understand its purpose and you are willing to participate in order to evaluate if you could safely participate in the study.

Do you have any further questions related to the study or related this telephone interview?

Will you allow me to proceed with the interview questions and to document your answers?

IRB Number: «ID»

Date Approved «ApprovalDate»



IRB Number: «ID»

Date Approved «ApprovalDate»



Changing What's Possible